CLINICAL TRIAL: NCT03210701
Title: A New APPROACH to HIV Testing: Adaptation of POCT for Pharmacies to Reduce Risk and Optimize Access to Care in HIV - A Type II Hybrid Implementation-Effectiveness Study
Brief Title: A New APPROACH to HIV Testing: Adaptation of POCT for Pharmacies to Reduce Risk and Optimize Access to Care in HIV
Acronym: APPROACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Deborah Kelly, Associate Professor and Special Advisor of Innovation, Memorial University of Newfoundland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HREB-2016.178
Record Dates: First submitted 2017-06-29; First posted 2017-07-07 (Actual); Results first posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: HIV Infections
Keywords: pharmacy; pharmacist; POCT; Implementation science
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients requesting a HIV screening test (Other)
  Interventions: Other: A HIV POCT program adapted for & provided by community pharmacists

INTERVENTIONS:
Other: A HIV POCT program adapted for & provided by community pharmacists — Using a Type II hybrid Implementation-Effectiveness study design investigators will assess the implementation and effectiveness of a multi-faceted, integrated, contextualized model of HIV POCT in pharmacies in urban and rural settings in NL and AB, Canada. This design will be flexible, responsive and capable of capturing changing elements at multiple points in time. A mixed methods approach will be used to assess Implementation and Effectiveness aims.

SUMMARY:
An estimated 21% of Canadians with HIV are unaware of their infection. There is a need to improve access to HIV testing to detect infections earlier so individuals can access care early and take steps to prevent transmission to others. Barriers to HIV testing include limited access or reluctance to go to traditional testing sites (doctor's offices and sexually transmitted infection clinics), and the lengthy wait time to receive test results from standard laboratory-based HIV testing (usually 1-2 weeks). These deterrents are particularly significant for those at highest risk of infection, who may be socially marginalized or stigmatized. In rural areas, HIV testing may only be available through doctor's offices and hospitals, yet many Canadians do not have access to a family physician. Pharmacists are among the most trusted and accessible healthcare providers, and are well positioned to improve access to HIV testing. Point of care tests for HIV are easy to administer and results are available within minutes, making them ideal for use in the community pharmacy setting. Point of care testing (POCT) by pharmacists can ensure individuals receive their test results, and facilitate timely linkages to care and treatment. This adaptation grant will look at factors influencing the acceptability and feasibility of pharmacist-provided rapid POCT for HIV in two Canadian provinces, including pharmacies in both urban and rural areas. The effectiveness of pharmacist-delivered POCT will be considered from a variety of perspectives including people living with or at risk of HIV, as well as pharmacists as the service providers.

DETAILED DESCRIPTION:
Background: There is a need to improve access to HIV testing to detect infections earlier so individuals can access care and prevent transmission. Barriers to testing include limited access or reluctance to go to traditional testing sites, and the lengthy wait time to receive results. Pharmacists are trusted, accessible health providers and are well positioned to offer HIV testing. Point of care tests (POCT) for HIV are easy to administer and results available within minutes, making them ideal for use in the pharmacy setting. HIV POCT may overcome barriers to standard testing for those at high risk and in healthcare resource-limited settings. Preliminary data suggest pharmacist-administered POCT can reach those who have never had an HIV test. Implementation and effectiveness of pharmacist-delivered POCT is the focus of this study. Study goals: To determine whether a multi-faceted HIV POCT program adapted for community pharmacies in two Canadian provinces is acceptable, feasible and effective in reaching those at high risk and those who have never been tested. Implementation and effectiveness of an integrated, contextualized model of HIV POCT in urban and rural pharmacies in Newfoundland (NL) and Alberta (AB) will be assessed. Participant characteristics, responses to satisfaction measures on the participant questionnaire, and pharmacist time to offer HIV POCT were analyzed using descriptive statistics. Pre-testing questionnaire data was used to calculate a Denver HIV Risk Score for each participant, as a means to predict their probability of having an undiagnosed HIV infection. ANOVA was used to assess differences in participants' Denver HIV Risk Scores between provinces, and urban versus rural testing sites, and multivariate analysis of variance (MANOVA) was used to assess differences in participant satisfaction with the testing experience based on province, urban/rural testing site, sex, and history of prior HIV testing. Fisher's Exact tests were used to assess whether history of prior HIV testing depended on province or urban/rural centre for testing. Qualitative data were analysed using a thematic analysis approach. Interview transcripts and extensive field notes were included for analysis from the participant interviews and pharmacist focus groups. Transcripts from participant interviews were coded using an open or emergent scheme where codes were developed and modified throughout the coding process. Descriptive codes were assigned to identify recurring concepts, and sub-themes were then identified and. Themes from the pharmacist focus groups were considered according to the Capability, Opportunity, Motivation, Behaviour (COM-B) model to understand behaviour change, which considers opportunities and challenges in the context of professional capability, opportunity, and motivation to offer the HIV POCT program. Impact: This study will inform further modifications to the pharmacy HIV POCT model to optimize effectiveness and increase scalability prior to full adoption and implementation. This will form the basis for a subsequent grant application. Knowledge gained can be used to scale up effective testing programs to increase the number of high risk individuals getting tested. The pharmacy is a novel venue to offer HIV testing, and if successful could be a widely accessible option applicable to other provinces and other countries. This study will provide proof of concept for pharmacy based POCT for other sexually transmitted and blood-borne infections (STBBI) (once tests become available) and successful implementation may also lead to pharmacist-delivered pre-exposure prophylaxis (PrEP) programs, to further reduce HIV infection rates.

ELIGIBILITY:
Inclusion Criteria:

* Consistent with current testing guidelines and the National HIV POCT Action Plan HIV testing will be offered to anyone age 18+ who requests a test and is not known to be HIV+.

Exclusion Criteria:

* Anyone unwilling to sign the consent form will be unable to participate in the study or receive HIV POCT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- School of Pharmacy, Memorial University, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kelly DV, Kielly J, Hughes C, Gahagan J, Asghari S, Hancock S, Burt K, Smyczek P, Charlton C, Nguyen H. Expanding access to HIV testing through Canadian community pharmacies: findings from the APPROACH study. BMC Public Health. 2020 May 7;20(1):639. doi: 10.1186/s12889-020-08719-0. PMID 32380978
- [Derived] Kielly J, Kelly DV, Hughes C, Day K, Hancock S, Asghari S, Gahagan J, Marra C, Nguyen H. Adaptation of POCT for pharmacies to reduce risk and optimize access to care in HIV, the APPROACH study protocol: examining acceptability and feasibility. Pilot Feasibility Stud. 2018 Feb 27;4:59. doi: 10.1186/s40814-018-0252-1. eCollection 2018. PMID 30788134

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Participants: Patients requesting a rapid HIV test at a community pharmacy study site.
Period: Overall Study
Arm/Group | Study Participants
Started | 123
Completed | 123
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Participants
Number analyzed (Participants) | 123
Age, Continuous [Mean (Full Range); unit: years] | 34.8 [18 to 97]
Sex/Gender, Customized [Number; unit: participants]
  Male | 93
  Female | 28
  Trans person | 0
  Other | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 98
  African, Caribbean or Black | 8
  Indigenous | 2
  Asian | 12
  Other | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Canada: Urban | 112
  Canada: Rural | 11
Relationship status [Count of Participants; unit: Participants]
  Single | 42
  Casually Dating | 39
  Married, Common-Law or Committed | 34
  Separted, divorced, widowed (SDW) | 6
  SDW and Casually Dating | 2
Employment Status [Count of Participants; unit: Participants]
  Full time | 76
  Part time | 4
  Student | 17
  Retired or on Disability | 9
  Not Employed | 12
  working and student | 4
  Other | 1
Highest level of education [Count of Participants; unit: Participants]
  Some high school | 2
  High school diploma or equivalent | 25
  Some university or college | 21
  Trade or technical school diploma | 30
  University degree | 45
Annual Income [Count of Participants; unit: Participants]
  <$20K | 32
  $20 - $39,999 | 25
  $40 - $59,999 | 26
  $60 - $79,999 | 11
  $80 - $99,999 | 14
  >$100K | 15
Tested for HIV previously [Count of Participants; unit: Participants]
  Tested previously | 86
  Not tested previously | 33
  Unsure | 2
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Patients Requesting a Rapid HIV Test at a Community Pharmacy Study Site
Description: Number of patients who presented to a community pharmacy test site and requested a rapid HIV test.
Time Frame: Collected at the end of the study period (6-8 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Study Participants
Number analyzed (Participants) | 123
Participants | 123

2. Primary Outcome: Number of Reactive Test Results
Description: Number of patients who requested a rapid HIV test at a community pharmacy and received a reactive test result
Time Frame: Collected at the end of the study period (6-8 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Study Participants
Number analyzed (Participants) | 123
Participants | 1

3. Primary Outcome: Total Time Required for the HIV Testing Process
Description: This was the time of the total patient pharmacist interaction, which began with the pharmacist explaining the study and ended with referring the patient for additional sexually transmitted blood borne infections (STBBI) counselling. The entire testing process included time spent explaining the study and consenting the participant, providing pre-test counselling, administering the test and explaining the result, post-test counselling, and referring the participant for additional STBBI testing as indicated.
Time Frame: From time of participant consenting through to providing pre-test counseling, administering the test & explaining the result, post-test counseling, & referring the participant for additional STBBI testing as indicated, 30-40 minutes on average
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Study Participants
Number analyzed (Participants) | 123
Minutes | 30.4 (6.95)

4. Primary Outcome: Participant Satisfaction With Testing Experience
Description: Once the testing was completed (see Outcome 3) prior to leaving, participants were asked to complete a de-identified, blinded questionnaire which assessed perception of the testing experience including factors that influenced their decision to be tested at the pharmacy & whether they would have sought HIV testing elsewhere if not at the pharmacy.
  Information was captured using a percentage continuous response scale from 0 to 100%. Participants were instructed to answer the questions by marking an "x" on the line at the point which represented their experience. For example, in response to the question "How likely are you to buy a lottery ticket today?", the participant was instructed that if they were 50% certain, they would mark an "x" at the 50% notch on the line.
  Questions were positively worded, with higher scores indicating higher agreement.
  Not all patients answered all questions; reported data is based on the number of respondents for each question.
Time Frame: Completed immediately after each individual participants testing process was completed, approximately 10 minutes on average
Population: Percentage continuous response scale (0-100)
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Study Participants
Number analyzed (Participants) | 123
score on a scale
  Comfort with testing at pharmacy: number analyzed (Participants) | 121
  Comfort with testing at pharmacy | 88.66 [0 to 100]
  Confidence PhC did a good job administering test: number analyzed (Participants) | 122
  Confidence PhC did a good job administering test | 96.93 [0 to 100]
  Likelihood to get tested for other STBBI: number analyzed (Participants) | 121
  Likelihood to get tested for other STBBI | 83.14 [0 to 100]
  Importance of privacy at pharmacy site: number analyzed (Participants) | 120
  Importance of privacy at pharmacy site | 89.42 [0 to 100]
  Importance of finger prick blood sample: number analyzed (Participants) | 120
  Importance of finger prick blood sample | 80.35 [0 to 100]
  Importance of immediate test results: number analyzed (Participants) | 120
  Importance of immediate test results | 94.87 [0 to 100]
  Importance of private room for testing and consult: number analyzed (Participants) | 120
  Importance of private room for testing and consult | 94.87 [0 to 100]
  Importance of free testing: number analyzed (Participants) | 121
  Importance of free testing | 88.78 [0 to 100]
  Imporatance of not needing an appointment: number analyzed (Participants) | 88
  Imporatance of not needing an appointment | 91.22 [0 to 100]
  Willingness to pay for testing: number analyzed (Participants) | 122
  Willingness to pay for testing | 78.69 [0 to 100]
  Should HIV testing be offered at pharmacies: number analyzed (Participants) | 122
  Should HIV testing be offered at pharmacies | 99.2 [0 to 100]

5. Primary Outcome: Participants Self-identified HIV Risk Behaviours
Description: Prior to initiating the testing process participants were asked to complete a de-identified, blinded questionnaire that included demographic data (age, gender, ethnicity, relationship status, highest education attained, and income level) as well as information about HIV risk factors and previous HIV testing history.
  Pre-testing questionnaire data on HIV risk factors was used to calculate a Denver HIV Risk Score (www.denverptc.org/resource.php?id=33) for each participant, as a means to predict their probability of having an undiagnosed HIV infection. Patients who score 30 points or greater on the Denver HIV Risk Score are considered at increased risk of undiagnosed HIV infection and should be offered routine screening.
  Not all patients answered all questions; numbers of respondents for each question is provided.
Time Frame: Immediately prior to testing process, participant completed the survey, approximately 5 - 10 minutes on average
Population: Not all patients answered all questions; numbers of respondents for each question is provided.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Participants
Number analyzed (Participants) | 123
Participants
  Men who have sex with men: number analyzed (Participants) | 119
  Men who have sex with men | 56
  History of IV drug use: number analyzed (Participants) | 118
  History of IV drug use | 6
  Previously exchanged sex for money or drugs: number analyzed (Participants) | 118
  Previously exchanged sex for money or drugs | 8
  Prior blood transfusion: number analyzed (Participants) | 118
  Prior blood transfusion | 2
  Denver HIV risk score >/= 30: number analyzed (Participants) | 118
  Denver HIV risk score >/= 30 | 89

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Study Participants
All-Cause Mortality (participants affected / at risk) | 0/123
Serious Adverse Events (participants affected / at risk) | 0/123
Other Adverse Events (participants affected / at risk) | 0/123

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-29): https://cdn.clinicaltrials.gov/large-docs/01/NCT03210701/Prot_SAP_000.pdf